CLINICAL TRIAL: NCT02545582
Title: VITARIA Registry Study
Status: Suspended | Type: Observational
Why Stopped: Sponsor decision
Sponsor: Cyberonics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: C-05
Record Dates: First submitted 2015-09-08; First posted 2015-09-10 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2016-03

CONDITIONS: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Therapy: Heart failure patients implanted with the VITARIA system
  Interventions: Device: VITARIA System

INTERVENTIONS:
Device: VITARIA System — Implantable vagus nerve stimulator

SUMMARY:
This registry will observe patients with symptomatic heart failure with implantable vagus nerve stimulation to provide insights into safety and efficacy during clinical routine.

DETAILED DESCRIPTION:
Observational prospective clinical registry in patients with symptomatic heart failure and implanted with the VITARIA System. Assessments will be made during 12 months of post-titration chronic stimulation. The registry will collect patient- and device follow-up data in clinical routine practice at baseline, 3, 6 and 12 months. Clinical routine safety of the therapy will be assessed by the incidence of procedure and device-related events. Clinical routine efficacy will be assessed by changes in cardiac function and heart failure symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and capable of providing informed consent according to national data privacy regulations
2. Patients with NYHA class II/III
3. LVEF≤40% by imaging method such as echocardiography, radionuclide angiography, left ventriculography, or cardiac magnetic resonance imaging, documented less than 12 weeks before implantation of VITARIA system
4. Receiving optimal pharmacological heart failure therapy for at least 3 months
5. Recent implantation of the VITARIA system, prior to device activation

Exclusion Criteria:

1. Hospitalization for heart failure and/or required the use of Heart Failure intravenous therapy in the past 30 days
2. Severe mitral and/or any aortic valve dysfunction
3. History of acute coronary syndrome (ACS) in the past 90 days
4. Stroke or transient ischemic attack (TIA) in the past 90 days
5. Coronary Artery Bypass Surgery (CABG) in the past 90 days
6. PCI in the past 90 days
7. Surgery for Valve replacement (Aortic or mitral valve) in the past 90 days
8. Left ventricular end diastolic diameter (LVEDD) > 80 mm
9. Patients who have had a cardiac resynchronization therapy (CRT) device implanted and have been actively treated with CRT for < 12 months
10. Patients that are scheduled for CRT
11. Patients who are listed for heart transplant or expected to be candidates for heart transplant
12. Patients on hemodialysis or peritoneal dialysis
13. Patients with diabetes (type I or type II) that is being medically treated for autonomic or sensory neuropathy, or measured hemoglobin A1c (HbA1c) above 8.0% in the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic heart failure, NYHA class II/III with LVEF≤40%
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-08; Primary Completion 2018-08 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 12 months
  Serious and non-serious adverse events, according to ISO 14155
LVEF | 12 months
  Left ventricular ejection fraction

SECONDARY OUTCOMES:
LVESV | 12 months
  Left ventricular end-systolic volume
LVESV Index | 12 months
  Left ventricular end-systolic volume index
NYHA Class | 12 months
  New York Heart Association classification
Quality of Life | 12 months
  Minnesota Living with Heart Failure Questionnaire
Heart Rate | 12 months
  Mean heart rate, 24-hour ambulatory ECG
Heart Rate Variability | 12 months
  SDNN, 24-hour ambulatory ECG

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Klein, MD, Principal Investigator — CRI GmbH
Locations (1):
- CRI GmbH, Munich, Germany